CLINICAL TRIAL: NCT02009241
Title: Evaluation of the Impact of a Pulmonary Rehabilitation Program on Exercise Capacity in Patients With Lymphangioleiomyomatosis
Brief Title: Pulmonary Rehabilitation in Lymphangioleiomyomatosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Mariana Sponholz Araujo, Postgraduate student, University of Sao Paulo General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22729413.6.0000.0068
Record Dates: First submitted 2013-12-04; First posted 2013-12-11 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Lymphangioleiomyomatosis
Keywords: Lymphangioleiomyomatosis; Rehabilitation; Exercise
MeSH Terms: conditions — Lymphangioleiomyomatosis; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pulmonary Rehabilitation (Active Comparator): The intervention group will perform a 12 week pulmonary rehabilitation program consisting of 30 minutes of treadmill aerobic exercise training and 30 minutes of muscle strength training.
  Interventions: Other: Pulmonary Rehabilitation
- Control (No Intervention)

INTERVENTIONS:
Other: Pulmonary Rehabilitation
  Arms: Pulmonary Rehabilitation

SUMMARY:
Lymphangioleiomyomatosis (LAM) is a rare disease in which reduced exercise capacity is frequently present. The mechanisms applied are airflow obstruction, abnormal diffusion capacity and dynamic hyperinflation (DH).

Pulmonary rehabilitation (PR) has proved benefit in improving exercise tolerance, dyspnea, and quality of life in chronic obstructive pulmonary disease. There are no studies evaluating the impact of PR in patients with LAM.

The hypothesis under study is that PR determine improvement in exercise capacity, dyspnea, quality of life, muscle force, functional limitation and DH in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of lymphangioleiomyomatosis established by tissue biopsy and / or a combination of history and high-resolution computed tomography scanning
* Clinical stability, defined as no exacerbations or hospitalizations related to the underlying disease for a minimum of 6 weeks and no change in the treatment regimen in the last 3 months
* Low level of physical activity, defined as patients who walk less than 10 thousand daily steps and / or are not performing regular physical activity for at least 4 months before the start of rehabilitation
* Signature of the free, prior and informed consent for participation in the study

Exclusion Criteria:

* Lung transplant recipients
* Musculoskeletal disorders that would prevent the patient from performing exercise training
* Severe (NYHA IV) or uncontrolled heart disease

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-11; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Endurance time during constant work rate cycle ergometry | 12 weeks

SECONDARY OUTCOMES:
Peak oxygen consumption (VO2 peak) during constant work rate cycle ergometry | 12 weeks
Dynamic hyperinflation and ventilatory parameters during constant work rate cycle ergometry | 12 weeks
Dyspnea and fatigue in the lower limbs during constant work rate cycle ergometry | 12 weeks
Dyspnea and functional disability related to daily life activities | 12 weeks
  The Modified Medical Research Council Dyspnea Scale (mMRC) and Baseline Dyspnea Index (BDI) will be evaluated pre - and post - intervention
Health factors related to quality of life | 12 weeks
  St. George's Respiratory Questionnaire (SGRQ) pre - and post - intervention
Anxiety and depression | 12 weeks
  Hospital Anxiety and Depression Scale (HADS) performed pre - and post - intervention
Daily physical activity | 12 weeks
  Evaluated using a pedometer for one week pre - and post - intervention
Changes in six minute walking distance and in desaturation - distance ratio (DDR) | 12 weeks
Changes in pulmonary function parameters | 12 weeks
Changes in peripheral muscle force | 12 weeks
  Using one repetition maximum (1 RM) pre - and post - intervention

CONTACTS AND LOCATIONS:
Overall Officials: Mariana S Araujo, MD, Principal Investigator — Pulmonary Division, Heart Institute (InCor), University of Sao Paulo Medical School; Carlos RR Carvalho, PhD, Principal Investigator — Pulmonary Division, Heart Institute (InCor), University of Sao Paulo Medical School
Locations (1):
- Pulmonary Division, Heart Institute (InCor), University of Sao Paulo Medical School, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Araujo MS, Baldi BG, Freitas CS, Albuquerque AL, Marques da Silva CC, Kairalla RA, Carvalho CR, Carvalho CR. Pulmonary rehabilitation in lymphangioleiomyomatosis: a controlled clinical trial. Eur Respir J. 2016 May;47(5):1452-60. doi: 10.1183/13993003.01683-2015. Epub 2016 Feb 25. PMID 26917604